CLINICAL TRIAL: NCT00644046
Title: Chronic Kidney Disease Prevention of An-Lo District, Keelung.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, iwenwu, Attending Physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IWW-0001; CGMH-IRB-96-0408B
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease; Death
Keywords: Chronic Kidney Disease; Prevention; Cardiovascular disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Death; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Chronic kidney disease patient with standardized nephrology care
- 2 (Active Comparator): chronic kidney disease patient with multidisciplinary predialysis care
  Interventions: Behavioral: multidisciplinary predialysis education

INTERVENTIONS:
Behavioral: multidisciplinary predialysis education — teaching of renal knowledges, dietary support and recall of period medical visits
  Other Names: MPE
  Arms: 2

SUMMARY:
The prevalence and the incidence of the end-stage renal disease (ESRD) are extremely high in Taiwan (1, 2). More than 45,000 patients are under renal replacement therapy in the year 2004 (2). The disease had not only caused a significant impact in personal life, but also a great burden on social security and government-run health insurance. However, despite this high prevalence, the awareness of chronic kidney disease (CKD) in general population remains low (3, 4). The patients always come out too late for the intervention to slow down the progression of renal failure. Furthermore, most of them are not well prepared for the renal replacement therapy. The facts result in high mortality and morbidity in this specific population (5). It is mandatory to screen out and treat these patients early enough. However, these patients are deep into the community as the asymptomatic nature of CKD.

The major purpose of the study is to screen the community for the early CKD and provide the appropriate intervention at time. The study will collect the characteristic demographic epidemiological data and find out risk factors for CKD of this geographic area, provide multidisciplinary education of CKD and establish timely referral for appropriate nephrologist care for treatment and monitoring of complications.

DETAILED DESCRIPTION:
The project will be last for 3 years. We will start to screen the patients within the community to identify the CKD population. This population will randomized into two group (one group with standard nephrologist care and another group with standard nephrologist care plus multidisciplinary CKD education) to evaluate the effectiveness of CKD education on the progression of renal function. The primary end-point will be the doubling tine estimated GFR, development of end-stage renal disease and all cause mortality. The non-CKD group of community will also follow up for urine and blood test for renal function, to determine the incidence and risk factors of new-onset renal disease. The accomplishment of this study will retard renal progression, improve community health and establish a model in preventing the chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* All CKD patients older than 18 y/o.

Exclusion Criteria:

* Refusal to participate in the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
reduction of estimated glomerular filtration rate by 50 % | 1 year

SECONDARY OUTCOMES:
death | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Iwen Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Division of Nephrology, Keelung, Taiwan

REFERENCES:
- [Background] Devins GM, Mendelssohn DC, Barre PE, Binik YM. Predialysis psychoeducational intervention and coping styles influence time to dialysis in chronic kidney disease. Am J Kidney Dis. 2003 Oct;42(4):693-703. doi: 10.1016/s0272-6386(03)00835-7. PMID 14520619
- [Background] Hsu CC, Hwang SJ, Wen CP, Chang HY, Chen T, Shiu RS, Horng SS, Chang YK, Yang WC. High prevalence and low awareness of CKD in Taiwan: a study on the relationship between serum creatinine and awareness from a nationally representative survey. Am J Kidney Dis. 2006 Nov;48(5):727-38. doi: 10.1053/j.ajkd.2006.07.018. PMID 17059992
- [Derived] Yu YJ, Wu IW, Huang CY, Hsu KH, Lee CC, Sun CY, Hsu HJ, Wu MS. Multidisciplinary predialysis education reduced the inpatient and total medical costs of the first 6 months of dialysis in incident hemodialysis patients. PLoS One. 2014 Nov 14;9(11):e112820. doi: 10.1371/journal.pone.0112820. eCollection 2014. PMID 25398129